CLINICAL TRIAL: NCT03050060
Title: ImmunoRad: Stratified Phase II Trial of Image Guided Hypofractionated Radiotherapy With Concurrent Nelfinavir and Immunotherapy in Advanced Melanoma, Lung Cancer, and Renal Cell Carcinoma
Brief Title: Image Guided Hypofractionated Radiation Therapy, Nelfinavir Mesylate, Pembrolizumab, Nivolumab and Atezolizumab in Treating Patients With Advanced Melanoma, Lung, or Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow accrual
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ramesh Rengan, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9712; NCI-2016-01816 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9712 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG3117000 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Results first posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-05

CONDITIONS: Metastatic Kidney Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Stage IV Cutaneous Melanoma AJCC v6 and v7; Stage IV Renal Cell Cancer AJCC v7; Stage IV Lung Non-Small Cell Cancer AJCC v7
Keywords: Kidney; Lung; Melanoma, Skin
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Melanoma | interventions — atezolizumab; Radiation Dose Hypofractionation; Radiation; Nelfinavir; Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nelfinavir, immunotherapy, radiation therapy) (Experimental): Beginning 7-14 days prior to start of pembrolizumab, nivolumab, or atezolizumab, patients receive nelfinavir mesylate PO BID on days 1-7 or 1-14 (dependent upon when treatment is started) up to 11-12 weeks. Patients also receive pembrolizumab, nivolumab or atezolizumab IV over 30-60 minutes on day 1. Cycles repeat every 21-28 days in the absence of disease progression or unacceptable toxicity. Patients then undergo hypofractionated radiation therapy over 3-14 days starting after cycle 1 and before cycle 3 of pembrolizumab, nivolumab or atezolizumab. The study will exclude irradiation of liver metastases as an added precaution.
  Interventions: Drug: Atezolizumab; Radiation: Hypofractionated Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: Nelfinavir Mesylate; Biological: Nivolumab; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated Radiotherapy; hypofractionation; Radiation, Hypofractionated
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nelfinavir Mesylate — Given PO
  Other Names: AG1343; Viracept
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well image guided hypofractionated radiation therapy works with nelfinavir mesylate, pembrolizumab, nivolumab, and atezolizumab in treating patients with melanoma, lung cancer, or kidney cancer that has spread (advanced). Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects. Nelfinavir mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as pembrolizumab, nivolumab and atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving hypofractionated radiation therapy, nelfinavir mesylate, pembrolizumab, nivolumab and atezolizumab may work better in treating patients with melanoma, lung, or kidney cancer.

DETAILED DESCRIPTION:
OUTLINE:

Beginning 7-14 days prior to start of pembrolizumab, nivolumab, or atezolizumab, patients receive nelfinavir mesylate orally (PO) twice daily (BID) on days 1-7 or 1-14 (dependent upon when treatment is started) up to 11-12 weeks. Patients also receive pembrolizumab, nivolumab or atezolizumab intravenously (IV) over 30-60 minutes on day 1. Cycles repeat every 21-28 days in the absence of disease progression or unacceptable toxicity. Patients then undergo hypofractionated radiation therapy over 3-14 days starting after cycle 1 and before cycle 3 of pembrolizumab, nivolumab or atezolizumab.

After completion of study treatment, patients are followed up at 30 days and then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Disease eligibility and stage

  * Histologically confirmed diagnosis of melanoma, non-small cell lung cancer (NSCLC), or renal carcinoma
  * Previously treated or previously untreated stage IV melanoma, stage IV or recurrent lung cancer, and metastatic renal cancer by American Joint Committee on Cancer (AJCC) staging criteria
  * Presence of a lesion that is suitable for hypofractionated radiotherapy
* Subjects must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria independent of the lesion to be irradiated. Prior checkpoint inhibitor immunotherapy or chemotherapy is allowed as long as the last dose was received > 14 days prior to enrollment
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Acceptable marrow function and hematologic indices for PD1/PDL1 immune checkpoint inhibitor and nelfinavir as per standard of care
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Subjects who have had immunotherapy, chemotherapy, or radiation therapy within 14 days (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Subjects may not be receiving other investigational agents
* Patients with untreated/active brain metastases as documented by computed tomography (CT) or magnetic resonance imaging (MRI) within 2 months of study enrollment; by active brain metastases - we mean - actively symptomatic brain metastases requiring steroids
* Allergy or intolerance to nelfinavir or selected PD1/PDL1 immune checkpoint inhibitor
* Patients requiring steroids or other immunosuppressive therapy; low-dose or topical steroids are allowable if being used as replacement therapy
* Patients receiving anti-retroviral therapy or other agents that are contra-indicated with nelfinavir due to drug-drug interactions*
* Pregnant or lactating patients
* Prior radiation that precludes delivery of hypofractionated radiotherapy

  * *For a study regarding the safety and efficacy of high dose nelfinavir on patients with Kaposi's Sarcoma (KS), exclusion criteria included participants who were receiving any "strong inhibitors or inducers of cytochrome P450, family 3, subfamily A (CYP3A) or cytochrome P450, family 2, subfamily C, polypeptide 19 (2C19)"

Strong Inhibitors of CYP3A4:

* Antibiotics: clarithromycin, erythromycin, telithromycin, troleandomycin
* HIV: non-nucleoside reverse transcriptase inhibitors (delavirdine, nevirapine), protease inhibitors (ritonavir, indinavir, lopinavir/ritonavir, saquinavir), cobicistat-boosted antiretrovirals (e.g., elvitegravir); NOTE: Clinical trials have demonstrated that there are no clinically significant drug-drug interactions between nelfinavir and the following antiretrovirals: efavirenz (strong CYP3A4 inhibitor), etravirine (strong CYP3A4 inhibitor); therefore, these antiretrovirals will not be excluded. • Antifungals: itraconazole, ketoconazole, voriconazole, fluconazole, posaconazole
* Antidepressants: nefazodone
* Antidiuretic: conivaptan
* GI: cimetidine, aprepitant
* Hepatitis C: boceprevir, telaprevir
* Miscellaneous: seville oranges, grapefruit, or grapefruit juice and/or pomelos, star fruit, exotic citrus fruits, or grapefruit hybrids.

Strong Inducers of CYP3A4:

* Glucocorticoids: cortisone (> 50 mg), hydrocortisone (> 40 mg), prednisone (> 10 mg), methylprednisolone (> 8 mg), dexamethasone (> 1.5 mg)
* Anticonvulsants: phenytoin, carbamazepine, primidone, phenobarbital and other enzyme inducing anti-convulsant drugs (EIACD)
* Antibiotics: rifampin (rifampicin), rifabutin, rifapentine
* Miscellaneous: St. John's Wort, modafinil

Strong Inhibitors of CYP2C9:

• Antifungals: fluconazole; lists including medications and substances known or with the potential to interact with the CYP3A or 2C19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2020-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Rengan, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We consented 21 patients but 1 patient was not eligible. Therefore, there are only 20 patients in the number of participants.
Period: Overall Study
Arm/Group | Treatment (Nelfinavir, Immunotherapy, Radiation Therapy)
Started | 20
Completed | 5
Not Completed | 15
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 1
Not completed — Progression | 7

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nelfinavir, Immunotherapy, Radiation Therapy)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Will be determined by immune-related Response Evaluation Criteria in Solid Tumor 1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT Scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.",
Time Frame: Up to 6 months after initiating treatment
Population: All patients starting trial therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nelfinavir, Immunotherapy, Radiation Therapy)
Number analyzed (Participants) | 17
Participants | 2

2. Secondary Outcome: Overall Survival
Description: Any long term data in the medical record that showed survival was use to measure overall survival.
Time Frame: From start of study treatment to death due to any cause, assessed up to 2 years
Population: 2 Patients were lost to follow-up before 2 year mark, 1 patient passed away during treatment due to Myocardial infarction, so they were not considered in the OS data.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nelfinavir, Immunotherapy, Radiation Therapy)
Number analyzed (Participants) | 17
Participants
  OS after 2 years (Renal) | 2
  OS after 2 years (Melanoma) | 3
  Patient death occurred prior to 2 years | 12

3. Secondary Outcome: Progression-free Survival
Description: No RECIST measurable progression over the course of 2 years post-treatment. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From start of treatment to progression by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, symptomatic deterioration, or death due to any cause, assessed up to 2 years
Population: 2 participants were lost to follow-up before the 2-year mark.
  1 Patient passed away during treatment due to a myocardial infraction.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nelfinavir, Immunotherapy, Radiation Therapy)
Number analyzed (Participants) | 17
Participants | 2

4. Secondary Outcome: Number of Adverse Events
Description: Will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. All adverse events that were attributable to study intervention in 20 participants, and counted the frequency of severity levels in the participants.
Time Frame: Adverse events were assessed up to 6 months from start of study treatment and All Cause Mortality was assessed upto 2 years from start of study treatment.
Measure: Number; unit: Percentage of adverse events
Units Other Than Participants: Adverse Events
Arm/Group | Treatment (Nelfinavir, Immunotherapy, Radiation Therapy)
Number analyzed (Participants) | 20
Number analyzed (Adverse Events) | 83
Percentage of adverse events
  Percentage of mild adverse events | 59
  Percentage of Moderate Adverse Events | 23
  Percentage of Severe Adverse Events | 14.5
  Percentage of Life-Threatening Adverse Events | 3.5

5. Secondary Outcome: Immune Correlative Studies: Changes in T-cell Repertoire
Description: Changes in T-cell receptor diversity
Time Frame: Up to 6 months
Population: Bio-specimens have been collected and stored, and cannot be analyzed by a processing team due to COVID-19 staffing limitations.
Arm/Group | Treatment (Nelfinavir, Immunotherapy, Radiation Therapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events are assessed during study treatment and study follow-up until the patient is removed from study (15 patients study length is 6-8 weeks, 5 patients study length 6 months.). The overall survival outcome measure data was assessed up to 2 years.
Arm/Group | Treatment (Nelfinavir, Immunotherapy, Radiation Therapy)
All-Cause Mortality (participants affected / at risk) | 12/20
Serious Adverse Events (participants affected / at risk) | 10/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nelfinavir, Immunotherapy, Radiation Therapy) (N=20)
AST Increased (Hepatobiliary disorders) | 8 (8)
ALT increased (Hepatobiliary disorders) | 10 (10)
Alk phos increased (Hepatobiliary disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nelfinavir, Immunotherapy, Radiation Therapy) (N=20)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cognitive Disturbance (Psychiatric disorders) | 1 (1)
Congestion (General disorders) | 1 (1)
Creatinine increase (Investigations) | 1 (1)
Dermatitis Radiaiton (Skin and subcutaneous tissue disorders) | 1 (1)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flashing Lights (Eye disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Insomnia (Metabolism and nutrition disorders) | 1 (1)
Loss of appetite (Metabolism and nutrition disorders) | 1 (1)
Lymphedema (Blood and lymphatic system disorders) | 1
Malaise (General disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lipase increase (Investigations) | 1 (1)
Increased Serum Amylase (Investigations) | 1 (1)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Sleep apnea (General disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Glucose 149 (Investigations) | 1 (1)
Increased Alkaline Phosphate (Investigations) | 2 (2)
Increased Serum Bilirubin (Investigations) | 2 (2)
Dehydration (General disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Fever (General disorders) | 1 (2)
Hot Flashes (General disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (2)
Skin Itchiness (Skin and subcutaneous tissue disorders) | 2 (2)
Weight gain (Metabolism and nutrition disorders) | 2 (2)
Weight Loss (Metabolism and nutrition disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Chills (General disorders) | 3 (3)
Hyperglycemia (Investigations) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4)
Dry mouth (General disorders) | 3 (4)
Dysgeusia (Gastrointestinal disorders) | 3 (5)
Urinary frequency (Renal and urinary disorders) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Headache (General disorders) | 6 (7)
Increased AST (Investigations) | 6 (8)
Vomiting (Gastrointestinal disorders) | 5 (9)
Increased ALT (Investigations) | 7 (10)
Fatigue (General disorders) | 11 (15)
Nausea (Gastrointestinal disorders) | 10 (19)
Diarrhea (Gastrointestinal disorders) | 15 (24)
Pain (General disorders) | 13 (39)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT03050060/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT03050060/ICF_001.pdf